CLINICAL TRIAL: NCT05942404
Title: Investigation of the Effect of Preoperative Bowel Cleansing on Lipopolysaccharide Binding Protein, Brain-Derived Neurotrophic Factor and Tau Protein Levels and Their Relationship With Postoperative Cognitive Impairment
Brief Title: Investigation of the Effect of Preoperative Bowel Cleansing on Postoperative Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Ulgey, PROFESSOR DR, TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2022/785
Record Dates: First submitted 2023-06-14; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: POCD - Postoperative Cognitive Dysfunction; Mechanical Bowel Preparation
Keywords: POCD; TAU PROTEİN; BDNF; LBP
MeSH Terms: conditions — Postoperative Cognitive Complications; Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of no bowel preparation (No Intervention): none mechanical bowel preparation
- Group of bowel preparation (Active Comparator): mechanical bowel preparation
  Interventions: Procedure: mechanical bowel preparation

INTERVENTIONS:
Procedure: mechanical bowel preparation — mechanical bowel preparation before surgery
  Arms: Group of bowel preparation

SUMMARY:
Cognitive impairment has been reported up to 54 % after colorectal surgeries. Mechanical bowel cleansing means that a system called the second brain in the body, which includes a wide variety of genetic and neuronal structures, is damaged. 100 trillion microorganisms live in the human body. The largest contact area with the external environment in the body, is the gastrointestinal mucosa. Microorganisms in the gut contain 100 times more genes than the human genome. The GI mucosa contains more than 500 million neurons called the enteric nervous system. MBP is an application that disrupts the microbiota structure and causes dehydration and electrolyte imbalance. While the most serious indication for MBP is seen as infection and health of anastomosis, recent studies say that this is not the case, even that the deterioration of the microbiota content damages the mucosal barrier, predisposes to inflammation with the removal of beneficial microorganisms and impairs wound healing.

84 patients will be included in the study, divided into two groups. In each group, blood will be drawn to measure the levels of biomarkers determined before surgery and bowel cleansing, on the 15th postoperative day and on the 90th day. Simultaneously, psychometric tests will be performed to assess cognitive impairment.

DETAILED DESCRIPTION:
In this project, the effects of pre-surgical mechanical bowel preperation on lipopolysaccharide binding protein (LBP), brain-derived neurotrophic factor (BDNF) and Tau protein levels and their relationship with postoperative cognitive dysfunction (PKB) are investigated. 84 patients will be included in the study, divided into two groups. In each group, blood will be drawn to measure the levels of biomarkers determined before surgery and bowel cleansing, on the 15th postoperative day and on the 90th day, and will be studied with the ELISA method. Simultaneously, psychometric tests will be performed to assess cognitive impairment.

Postoperative cognitive impairment (PCI) is defined as deterioration and worsening of cognitive status that occurs after surgery and lasts more than 30 days and less than 12 months. Postoperative neurological diseases are an increasing research and curiosity in the world, and unfortunately, knowledge and experience on this subject are very limited. With the aging of the population worldwide and the increasing number of elderly patients requiring surgical intervention, the incidence of postoperative neurological complications is increasing. PCD increases mortality, causes serious economic losses, psychological and social problems in the society and the family. The most important reason in the pathophysiology of PCD is the inflammatory response secondary to surgical intervention.

Cognitive impairment has been reported up to 54 % after colorectal surgeries. In colorectal surgery, different from other major surgeries, bowel cleansing is performed. Mechanical bowel cleansing means that a system called the second brain in the body, which includes a wide variety of genetic and neuronal structures, is damaged. 100 trillion microorganisms live in the human body. Our system, which has the largest contact area with the external environment in the body, is the GIS mucosa. Microorganisms in the gut contain 100 times more genes than the human genome. The GI mucosa contains more than 500 million neurons called the enteric nervous system. Approximately 1012-13 microorganisms living in the GIS are in close relationship with this enteric nervous system with their genetic materials.

Many studies have shown that the microbiota-gut-brain connection is effective in the formation of neurodegenerative diseases. In animal studies, it has been shown that temporary changes in the microbiota affect the brain chemical structure and behavior of the animal. Recent studies show that the microbiota, which is an environmental factor, has important effects on the brain. In intestinal surgeries, mechanical bowel preperation (MBP) was performed, considering that the intestinal microbiota would prepare the ground for infection. In recent years, the question of whether MBP should be done has been seriously questioned. MBP is an application that disrupts the microbiota structure and causes dehydration and electrolyte imbalance. While the most serious indication for MBP is seen as infection and health of anastomosis, recent studies say that this is not the case, even that the deterioration of the microbiota content damages the mucosal barrier, predisposes to inflammation with the removal of beneficial microorganisms and impairs wound healing.

Prevention of PCD is very important. Because the development of PKD is an important indicator for the first year mortality in noncardiac surgeries. Patients with PCD at discharge die within 3 months. Patients with persistent PCD in the first 3 months postoperatively die within the first year.

Our aim in this study is to investigate the effectiveness of certain biomarkers and whether there is a relationship between their levels and the development of cognitive impairment in the postoperative period in order to evaluate the clinical reflections of the microbiota environment that has been intervened by performing MBT in colorectal surgeries that have never been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to participate in the study
* Patients undergoing elective colorectal surgery
* Patients who can read and write
* Patients whose hearing and sight are suitable for communication
* Patients whose general sociocultural status is sufficient to perform psychometric tests.

Exclusion Criteria:

* Patients with inflammatory bowel
* Patients with cerebrovascular disease
* Patients who require emergency surgery
* Patients who have had repetitive surgeries
* Patients with neurodegenerative disease
* Patients with severe and moderate dementia (MoCA test score 21 and below)
* Patients with a mini mental test below 24
* Patients with severe hearing and vision impairment
* Patients using antibiotics and probiotics
* Patients who take long-term steroid therapy (7 days or more)
* Patients receiving immunosuppressive therapy

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2023-07-22 (Estimated); Primary Completion 2024-07-21 (Estimated); Study Completion 2024-07-21 (Estimated)

PRIMARY OUTCOMES:
the incidence of postoperative cognitive disfunction | 3
  1st day before the operation, 15th day and 90th day after the operation the psychometric tests will be performed to evaluate POCD relevant biomarkers will also be measured